CLINICAL TRIAL: NCT04122248
Title: M6-C Artificial Cervical Disc IDE Post Approval Study
Brief Title: M6-C Post Approval Study (PAS)
Status: Active, not recruiting | Type: Observational
Sponsor: Spinal Kinetics (Industry)
Responsible Party: Sponsor
Organization: Orthofix Inc. (Industry)
Other Study IDs: CA-C004
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cervical Degenerative Disc Disease; Cervical Radiculopathy; Cervical Spinal Cord Compression; Cervical Disc Herniation
Keywords: artificial cervical disc arthroplasty
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- M6-C: Subjects treated with an M6-C device
  Interventions: Other: standard radiographic imaging; Device: cervical total disc replacement
- ACDF: Subjects treated with Anterior Cervical Discectomy and Fusion (ACDF)
  Interventions: Other: standard radiographic imaging

INTERVENTIONS:
Other: standard radiographic imaging — standard radiographic imaging
Device: cervical total disc replacement — Artificial disc replacement (ADR) in the cervical spine is a minimally invasive procedure that involves removing diseased disc tissue and replacing it with an artificial disc. The artificial disc is designed to preserve the spine's natural motion while remaining securely attached to the surrounding vertebral bones. The goal of ADR is to help preserve the motion of the cervical spine or spinal segment after surgery, which can improve the quality of life for patients.
  Other Names: cervical disc arthroplasty; cervical artificial disc replacement
  Groups: M6-C

SUMMARY:
The M6-C Post Approval Study is a long term follow-up study of subjects previously enrolled and treated in the M6-C Artificial Cervical Disc IDE Study.

DETAILED DESCRIPTION:
A prospective, concurrently controlled, multi-center pivotal study to evaluate the safety and effectiveness of the M6-C™ Artificial Cervical Disc compared to anterior cervical discectomy and fusion (ACDF) was performed in the United States under IDE #G050254. To fulfill the concurrent control design of the study, there were clinical sites that evaluated the safety and effectiveness of the M6-C™ Artificial Cervical Disc and there were other clinical sites that evaluated ACDF. Subjects in the study were treated between May 2014 and June 2016 and remain in follow-up. The M6-C™ Artificial Cervical Disc received FDA approval to market on February 6, 2019. As a condition of approval, the FDA requested that the sponsor perform a post market approval study (PAS). The subjects enrolled and remaining in the M6-C IDE pivotal study are the prospective patient population for the PAS.

ELIGIBILITY:
Inclusion Criteria:

* Since the subjects have already been screened as part of the IDE's pivotal study, and only subjects that participated in that study make up the subject cohort for this long-term follow-up study, there are no additional inclusion criteria

Exclusion Criteria:

* Subjects who were withdrawn or withdrew consent to participate in the investigation
* Subjects who do not consent to participate in long-term follow-up or provide personal contact information to the sponsor (solely for the purposes of tracking subjects to help ensure follow-up compliance)
* Patients with terminal failures (SSI or device- or procedure-related SAE) by Month 24 and all known patient deaths in the M6-C IDE study are excluded for enrollment into the PAS

Ages: 21 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for study enrollment will include subjects implanted in the M6-C™ IDE pivotal study
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall subject success | 10 year follow-up
  A study subject will be considered an overall success if he/she meets the following criteria:
  * No serious adverse event(s) classified as device or device procedure related (as determined by the CEC), and
  * No subsequent surgical procedure at the index level (including revision, removal, reoperation, or supplemental fixation), and
  * Maintenance or improvement in neurological function, and
  * Improvement on the NDI of at least 15 points.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | annually to 10 years
  The NDI is a patient reported outcome questionnaire for the measurement of pain and function related to cervical spine problems. A total NDI score is determined by adding the scores of the individual questions and dividing that total by the maximum possible score (i.e., 50 if all questions are answered) to yield a percentage. Therefore, the NDI score ranges from 0% to 100%. A lower score represents less pain and dysfunction.
Neck and arm pain | annually to 10 years
  A visual analogue scale is a patient reported outcome measure utilized to determine neck and arm pain on a zero to ten scale with zero being the least amount of pain and 10 the most possible pain.
SF-36 Health Survey | annually to 10 years
  The SF-36 is a patient reported outcome questionnaire to measure health-related Quality of Life. An increase in score from baseline represents an improvement in health.
Patient Satisfaction | annually to 10 years
  The following 5 point Likert Scale will be used to further assess subject satisfaction:
  1. How satisfied are you with the results of your surgery? Very Satisfied; Satisfied; Neutral; Unsatisfied; Very Unsatisfied
  2. All things considered, would you have the surgery again? Very likely; likely; not sure; Unlikely; Very Unlikely
  3. Would you recommend the surgery to a friend or family member? Very likely; likely; not sure; Unlikely; Very Unlikely
Odom's Criteria | annually to 10 years
  At the 5, 7 and 10 year follow-up visits, the Investigator will rate the clinical disposition of each study subject according to Odom's Criteria[18] as follows:
  Excellent: No symptoms related to cervical disease. Able to perform daily activities without limitations.
  Good: Moderate symptoms related to cervical disease. Able to perform daily activities without significant limitations.
  Satisfactory: Slight improvement is symptoms related to cervical disease. Significant limitations in daily activities.
  Poor: No improvement in, or aggravation of, symptoms related to cervical disease. Not able to perform daily activities.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Desert Institute for Spine Care, Phoenix, Arizona
  - The CORE Institute, Sun City West, Arizona
  - Spine MD, Beverly Hills, California
  - Memorial Orthopedic Surgical Group, Long Beach, California
  - Stanford University, Stanford, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - ClinTech Center for Spine, Johnstown, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Medstar Hospital/Georgetown University, Washington D.C., District of Columbia
  - Midwest Orthopedics, Chicago, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Spine Institute of Lousianna, Shreveport, Louisiana
  - HSS, New York, New York
  - Upstate Medical University, Syracuse, New York
  - CNSA, Charlotte, North Carolina
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - EmergeOrtho, Durham, North Carolina
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Center for Sports Medicine & Orthopedics, Chattanooga, Tennessee
  - Texas Back Institute, Plano, Texas
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No